CLINICAL TRIAL: NCT07026266
Title: Sponsored, Randomized, Double-blind, Single-center Study on the Effect of the Intake of a Calcium-bicarbonate Water (Lete) on Cholesterol Levels
Brief Title: Study on the Effect of the Intake of a Calcium-bicarbonate Water on Cholesterol Levels
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Società Generale delle Acque Minerali S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LDLete
Record Dates: First submitted 2025-05-30; First posted 2025-06-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-05

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Lete" group (Experimental): Calcium-bicarbonate mineral water "Lete"
  Interventions: Other: Water
- "Sorgesana" group (Active Comparator): Oligomineral water "Sorgesana"
  Interventions: Other: Water

INTERVENTIONS:
Other: Water — Calcium-bicarbonate mineral water "Lete"
  Arms: "Lete" group
Other: Water — Oligomineral water "Sorgesana"
  Arms: "Sorgesana" group

SUMMARY:
The goal of this study is to evaluate the hypolipidemic effect (reduction of Low Density Lipoprotein Cholesterol "LDL-C" values) of calcium-bicarbonate mineral water "Lete" (alkaline water, high in bicarbonate and calcium ions and low in sodium) compared to control oligomineral water "Sorgesana" on healthy volunteers

DETAILED DESCRIPTION:
This sponsored, monocentric and interventional study will consist of a screening visit, a baseline visit, a phone contact one month after the baseline visit and two follow-up visits in person, two and four months after the baseline visit. After signing the informed consent and verifying the eligibility criteria, 160 healthy subjects will be randomized in a 1:1 double-blind ratio to one of two study arms. During the baseline visit, informations regarding the patient's medical history, demographic, anthropometric and blood pressure data and concomitant medications will be collected and the patient will be asked to complete a questionnaire related to physical activity assessment and to undergo an evaluation test for proper nutrition. Then, a blood sample will be taken for hematochemical analysis to evaluate the study endpoints. Finally, during the two follow-up visits, treatment adherence will be assessed, a blood sample will be taken for hematochemical analysis and the patient will be asked to complete the questionnaire and to undergo the evaluation test for proper nutrition. Additionally, at the second follow-up visit, anthropometric and blood pressure data will be collected

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* age 18-60 years
* LDL-C values > 116 mg/dl
* not already being treated with cholesterol-lowering medications (e.g. statins, ezetimibe, monoclonal antibodies, bempedoic acid) and/or supplements (e.g. fermented red rice, coenzyme Q, folic acid, berberine, vitamin E, polyphenols from olive oil, etc.)

Exclusion Criteria:

* BMI < 20 and > 30 kg/m2
* diabetes mellitus
* arterial hypertension
* gastrointestinal (e.g. gastro-duodenal ulcer, ulcerative colitis, diverticulosis of the colon, etc.), liver or renal diseases
* familial hypercholesterolemia
* treatment with drugs that could influence lipid metabolism (estrogen replacement hormone therapy, corticosteroid therapy, insulin therapy)
* Consumers of fortified foods that could influence lipid metabolism (containing n-3 fatty acids or phytosterols)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Variation of LDL-C values after four months of treatment | Four months
  Variation of LDL-C values (in mg/dl) after four months of treatment with the calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water

SECONDARY OUTCOMES:
Variation of the anthropometric data of weight after two and four months of treatment | Four months
  Variation of the anthropometric data of weight (in kg) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the anthropometric data of Body Mass Index "BMI" after two and four months of treatment | Four months
  Variation of the anthropometric data of BMI (in kg/m^2) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the anthropometric data of abdominal circumference after two and four months of treatment | Four months
  Variation of the anthropometric data of abdominal circumference (in cm) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of blood pressure values after two and four months of treatment | Four months
  Variation of blood pressure values (in mmHg) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of heart rate after two and four months of treatment | Four months
  Variation of heart rate (in bpm) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of LDL-C values after two and four months of treatment | Four months
  Variation of LDL-C values (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of total cholesterol after two and four months of treatment | Four months
  Variation of the parameters of total cholesterol (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of High Density Lipoprotein "HDL" cholesterol after two and four months of treatment | Four months
  Variation of the parameters of HDL cholesterol (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of triglycerides after two and four months of treatment | Four months
  Variation of the parameters of triglycerides (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of Lipoprotein a "Lp(a)" after two and four months of treatment | Four months
  Variation of the parameters of Lp(a) (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of Apolipoprotein B-100 after two and four months of treatment | Four months
  Variation of the parameters of Apolipoprotein B-100 (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of Apolipoprotein A1 after two and four months of treatment | Four months
  Variation of the parameters of Apolipoprotein A1 (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of creatinine after two and four months of treatment | Four months
  Variation of the parameters of creatinine (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of uric acid after two and four months of treatment | Four months
  Variation of the parameters of uric acid (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of blood glucose after two and four months of treatment | Four months
  Variation of the parameters of blood glucose (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of glycated hemoglobin "HbA1c" after two and four months of treatment | Four months
  Variation of the parameters of HbA1c (in %) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of ASpartate Transaminase "AST" after two and four months of treatment | Four months
  Variation of the parameters of AST (in U/l) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of ALanine Transaminase "ALT" after two and four months of treatment | Four months
  Variation of the parameters of ALT (in U/l) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of gamma-Glutamyl Transferase "gamma-GT" after two and four months of treatment | Four months
  Variation of the parameters of gamma-GT (in U/l) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of alkaline phosphatase after two and four months of treatment | Four months
  Variation of the parameters of alkaline phosphatase (in U/l) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of lipase after two and four months of treatment | Four months
  Variation of the parameters of lipase (in U/l) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of high sensitivity C-Reactive Protein "hs-CRP" after two and four months of treatment | Four months
  Variation of the parameters of hs-CRP (in mg/l) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of sodium after two and four months of treatment | Four months
  Variation of the parameters of sodium (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of magnesium after two and four months of treatment | Four months
  Variation of the parameters of magnesium (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of potassium after two and four months of treatment | Four months
  Variation of the parameters of potassium (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of calcium after two and four months of treatment | Four months
  Variation of the parameters of calcium (in mg/dl) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water
Variation of the parameters of Vitamin D after two and four months of treatment | Four months
  Variation of the parameters of Vitamin D (in nmol/l) after two and four months of treatment with calcium-bicarbonate water in relation to baseline, for comparison with the control oligomineral water

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Margonato, Principal Investigator — Hospital San Raffaele - Milano (Italy)
Locations (1):
- Hospital San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No